CLINICAL TRIAL: NCT06156241
Title: Long COVID: Cord Tissue-Derived Mesenchymal Stromal Cells for Persistent NeuroInflammatory Symptoms
Brief Title: Stem Cell Study for Long COVID-19 Neurological Symptoms
Acronym: COVID-19
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Charles Cox (Other)
Collaborators: CBR Systems, Inc. (Other)
Responsible Party: Sponsor-Investigator, Charles Cox, The George and Cynthia Mitchell Distinguished Chair in Neurosciences Director, Children's Program in Regenerative Medicine Professor, Departments of Surgery and Pediatric Surgery UTHealth, McGovern Medical School at Houston, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-xxxx
Record Dates: First submitted 2023-11-17; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: Post COVID-19 Neurological Injuries
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Non-Randomized, Phase 1/2a dose escalation using 4X10^6/kg, 6X10^6/kg and 8X10^6/kg and 10X10^10/kg cohorts of 3 patients using an adaptive Bayesian design based upon infusional toxicity/safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 4x10^6 Cells/kg Dose Group (Experimental): This is a adaptive Baysian dose escalation study. The first 3 subjects will receive one stem cell infusion of 4x10^6 Cells/kg. If no infusion related AE/SAE are found, the next cohort will receive the next highest stem cell dose.
  Interventions: Biological: Stem Cell
- 6x10^6 Cells/kg Dose Group (Experimental): The next cohort of 3 subjects will receive one stem cell infusion of 6x10^6 Cells/kg.
  If no infusion related AE/SAE are found, the next cohort will receive the next highest stem cell dose.
  Interventions: Biological: Stem Cell
- 8x10^6 Cells/kg Dose Group (Experimental): The next cohort of 3 subjects will receive one stem cell infusion of 8x10^6 Cells/kg.
  If no infusion related AE/SAE are found, the next cohort will receive the next highest stem cell dose.
  Interventions: Biological: Stem Cell
- 10x10^6 Cells/kg Dose Group (Experimental): The last cohort of 3 subjects will receive one infusion of 10x10^6 Cells/kg.
  Interventions: Biological: Stem Cell

INTERVENTIONS:
Biological: Stem Cell — Stem cells derived from human cord tissue.
  Other Names: Allogenic Human Cord Tissue Derived Mesenchymal Stromal Cells (hCTMSCs)

SUMMARY:
The purpose of this research study is to test the safety and benefit of a human cord blood derived stem cell infusion as a treatment for individuals with post COVID-19 neurological problems. Participants in the study will have 6 clinic visits over a 12 to 14 mo. period with each visit lasting 2 to 6 hours. Participants will receive 1 stem cell infusion at study visit #3. Participants will have a brain PET and MRI scan at the baseline and 6mo. post-infusion visits. Follow-up safety assessments will be conducted at 6mo. and 1yr. after the stem cell infusion.

DETAILED DESCRIPTION:
This is a non-randomized, Phase 1/2a dose escalation study using allogenic cord tissue MSC's in adults with chronic neurological symptoms following an acute COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 18 and 55 years of age.
2. Documented history of COVID-19 infection with resulting neurological sequela.
3. Post-Covid-19 Functional Status score of grades 3 or 4.
4. Chronic neurological symptoms defined as anxiety/depression, pain syndromes, sleep disorders, and /or memory disorders ("brain fog") persisting 6 months after an acute COVID-19 infection.
5. Ability to obtain consent from the subject.
6. Ability to communicate in English or Spanish (required for validated neurocognitive outcome testing).

Exclusion Criteria:

1. Known history of:

   1. intellectual deficiency or psychiatric conditions likely to invalidate our ability to assess changes in cognition or behavior,
   2. recently treated infection,
   3. renal disease or altered renal function (screening serum creatinine > 1.5 mg/dL),
   4. hepatic disease or altered liver function (screening SGPT > 150 U/L and/or T. Bilirubin >1.3 mg/dL),
   5. cancer,
   6. immunosuppression (screening WBC < 3, 000 cells/ml),
   7. HIV+,
   8. chemical or ETOH dependency that in the opinion of the investigator would preclude participation in the study,
   9. acute or chronic lung disease requiring significant medication/oxygen supplementation,
   10. bleeding disorders including immune-mediated heparin-induced thrombocytopenia,
   11. hypercoagulable disorders (Protein C, S, ATIII deficiencies), Factor V Leiden,
   12. known sensitivity to heparin, Lovenox, and pork products,
   13. individuals with mechanical prosthetic heart valves.
2. Pulse oximetry oxygen saturation <93% on room air.
3. Other acute or chronic medical conditions that, in the opinion of the investigator, may increase the risks associated with study participation.
4. For women of childbearing potential, a positive pregnancy test at the screening visit or, for both women and men, unwillingness to comply with acceptable methods of birth control during the study.
5. Previous or concurrent participation in an interventional drug or biological study.
6. Inability to undergo the diagnostic tests (PET/DT-MRI) or unwilling/unable to cooperate with the diagnostic tests and outcome assessments.
7. Unwilling or unable to return for follow-up study visits.
8. Prisoner/Incarcerated.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Determine the safety and establish the maximum tolerated dose (MTD) of allogenic human cord tissue derived MSCs (hCTMSCs) as determined by infusional toxicity of the cell product. | Assessed for the first 24 hours after each stem cell infusion.
  Physical Exam
Determine the safety and establish the maximum tolerated dose (MTD) of allogenic human cord tissue derived MSCs (hCTMSCs) as determined by infusional toxicity of the cell product. | Assessed for the first 24 hours after each stem cell infusion.
  Clinical Lab Assessments
Determine the safety and establish the maximum tolerated dose (MTD) of allogenic human cord tissue derived MSCs (hCTMSCs) as determined by infusional toxicity of the cell product. | Assessed for the first 24 hours after each stem cell infusion.
  Vital Signs
Determine the safety and establish the maximum tolerated dose (MTD) of allogenic human cord tissue derived MSCs (hCTMSCs) as determined by infusional toxicity of the cell product. | Assessed for the first 24 hours after each stem cell infusion.
  Subject Report of Adverse Event(s)

SECONDARY OUTCOMES:
Investigate if the hCTMSC infusions reduce the neuroinflammatory response following an acute COVID-19 infection as measured by the degree of microglial activation. | Baseline visit to 6 months post-infusion.
  Comparison of Brain PET Scan at baseline visit and at 6 months post-infusion.

OTHER OUTCOMES:
Obtain treatment effect estimates on the structural integrity of the corpus callosum measured by changes in fractional anisotropy (FA). | Baseline visit to 6 months post-infusion.
  Comparison of Brain DT-MRI at baseline visit and at 6 month post-infusion.
Obtain treatment effect estimates on the structural integrity of the corpus callosum measured by mean diffusivity (MD). MD is an inverse measure of membrane density, and is sensitive to edema and necrosis. | Baseline visit to 6 months post-infusion.
  Comparison of Brain DT-MRI at baseline visit and at 6 month post-infusion.
Obtain treatment effect estimates on the structural integrity of the corticospinal tracts measured by fractional anisotropy (FA). | Baseline visit to 6 months post-infusion.
  Comparison of Brain DT-MRI at baseline visit and at 6 month post-infusion.
Obtain treatment effect estimates on the structural integrity of the corticospinal tracts measured by mean diffusivity (MD). MD is an inverse measure of membrane density, and is sensitive to edema and necrosis. | Baseline visit to 6 months post-infusion.
  Comparison of Brain DT-MRI at baseline visit and at 6 month post-infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Cox, MD, Principal Investigator — The Univ. of Tx. Health Science Center- Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aiyegbusi OL, Hughes SE, Turner G, Rivera SC, McMullan C, Chandan JS, Haroon S, Price G, Davies EH, Nirantharakumar K, Sapey E, Calvert MJ; TLC Study Group. Symptoms, complications and management of long COVID: a review. J R Soc Med. 2021 Sep;114(9):428-442. doi: 10.1177/01410768211032850. Epub 2021 Jul 15. PMID 34265229
- [Result] Cha C, Baek G. Symptoms and management of long COVID: A scoping review. J Clin Nurs. 2024 Jan;33(1):11-28. doi: 10.1111/jocn.16150. Epub 2021 Dec 15. PMID 34913540
- [Result] Costas-Carrera A, Sanchez-Rodriguez MM, Canizares S, Ojeda A, Martin-Villalba I, Prime-Tous M, Rodriguez-Rey MA, Segu X, Valdesoiro-Pulido F, Borras R, Peri JM, Vieta E. Neuropsychological functioning in post-ICU patients after severe COVID-19 infection: The role of cognitive reserve. Brain Behav Immun Health. 2022 May;21:100425. doi: 10.1016/j.bbih.2022.100425. Epub 2022 Feb 7. PMID 35156065
- [Result] Davis HE, Assaf GS, McCorkell L, Wei H, Low RJ, Re'em Y, Redfield S, Austin JP, Akrami A. Characterizing long COVID in an international cohort: 7 months of symptoms and their impact. EClinicalMedicine. 2021 Aug;38:101019. doi: 10.1016/j.eclinm.2021.101019. Epub 2021 Jul 15. PMID 34308300
- [Result] Del Rio C, Collins LF, Malani P. Long-term Health Consequences of COVID-19. JAMA. 2020 Nov 3;324(17):1723-1724. doi: 10.1001/jama.2020.19719. No abstract available. PMID 33031513
- [Result] Doykov I, Hallqvist J, Gilmour KC, Grandjean L, Mills K, Heywood WE. 'The long tail of Covid-19' - The detection of a prolonged inflammatory response after a SARS-CoV-2 infection in asymptomatic and mildly affected patients. F1000Res. 2020 Nov 19;9:1349. doi: 10.12688/f1000research.27287.2. eCollection 2020. PMID 33391730
- [Result] Graham EL, Clark JR, Orban ZS, Lim PH, Szymanski AL, Taylor C, DiBiase RM, Jia DT, Balabanov R, Ho SU, Batra A, Liotta EM, Koralnik IJ. Persistent neurologic symptoms and cognitive dysfunction in non-hospitalized Covid-19 "long haulers". Ann Clin Transl Neurol. 2021 May;8(5):1073-1085. doi: 10.1002/acn3.51350. Epub 2021 Mar 30. PMID 33755344
- [Result] Hayes LD, Ingram J, Sculthorpe NF. More Than 100 Persistent Symptoms of SARS-CoV-2 (Long COVID): A Scoping Review. Front Med (Lausanne). 2021 Nov 1;8:750378. doi: 10.3389/fmed.2021.750378. eCollection 2021. PMID 34790680
- [Result] Higgins V, Sohaei D, Diamandis EP, Prassas I. COVID-19: from an acute to chronic disease? Potential long-term health consequences. Crit Rev Clin Lab Sci. 2021 Aug;58(5):297-310. doi: 10.1080/10408363.2020.1860895. Epub 2020 Dec 21. PMID 33347790
- [Result] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Result] Ikawa M, Lohith TG, Shrestha S, Telu S, Zoghbi SS, Castellano S, Taliani S, Da Settimo F, Fujita M, Pike VW, Innis RB; Biomarkers Consortium Radioligand Project Team. 11C-ER176, a Radioligand for 18-kDa Translocator Protein, Has Adequate Sensitivity to Robustly Image All Three Affinity Genotypes in Human Brain. J Nucl Med. 2017 Feb;58(2):320-325. doi: 10.2967/jnumed.116.178996. Epub 2016 Nov 17. PMID 27856631
- [Result] Kayaaslan B, Eser F, Kalem AK, Kaya G, Kaplan B, Kacar D, Hasanoglu I, Coskun B, Guner R. Post-COVID syndrome: A single-center questionnaire study on 1007 participants recovered from COVID-19. J Med Virol. 2021 Dec;93(12):6566-6574. doi: 10.1002/jmv.27198. Epub 2021 Jul 28. PMID 34255355
- [Result] Lemhofer C, Gutenbrunner C, Schiller J, Loudovici-Krug D, Best N, Bokel A, Sturm C. Assessment of rehabilitation needs in patients after COVID-19: Development of the COVID-19-rehabilitation needs survey. J Rehabil Med. 2021 Apr 27;53(4):jrm00183. doi: 10.2340/16501977-2818. PMID 33764478
- [Result] Mandal S, Barnett J, Brill SE, Brown JS, Denneny EK, Hare SS, Heightman M, Hillman TE, Jacob J, Jarvis HC, Lipman MCI, Naidu SB, Nair A, Porter JC, Tomlinson GS, Hurst JR; ARC Study Group. 'Long-COVID': a cross-sectional study of persisting symptoms, biomarker and imaging abnormalities following hospitalisation for COVID-19. Thorax. 2021 Apr;76(4):396-398. doi: 10.1136/thoraxjnl-2020-215818. Epub 2020 Nov 10. PMID 33172844
- [Result] Malik P, Patel U, Mehta D, Patel N, Kelkar R, Akrmah M, Gabrilove JL, Sacks H. Biomarkers and outcomes of COVID-19 hospitalisations: systematic review and meta-analysis. BMJ Evid Based Med. 2021 Jun;26(3):107-108. doi: 10.1136/bmjebm-2020-111536. Epub 2020 Sep 15. PMID 32934000
- [Result] O'Connor RJ, Preston N, Parkin A, Makower S, Ross D, Gee J, Halpin SJ, Horton M, Sivan M. The COVID-19 Yorkshire Rehabilitation Scale (C19-YRS): Application and psychometric analysis in a post-COVID-19 syndrome cohort. J Med Virol. 2022 Mar;94(3):1027-1034. doi: 10.1002/jmv.27415. Epub 2021 Nov 5. PMID 34676578
- [Result] Ogier M, Andeol G, Sagui E, Dal Bo G. How to detect and track chronic neurologic sequelae of COVID-19? Use of auditory brainstem responses and neuroimaging for long-term patient follow-up. Brain Behav Immun Health. 2020 May;5:100081. doi: 10.1016/j.bbih.2020.100081. Epub 2020 May 15. PMID 32427134
- [Result] Paterson RW, Brown RL, Benjamin L, Nortley R, Wiethoff S, Bharucha T, Jayaseelan DL, Kumar G, Raftopoulos RE, Zambreanu L, Vivekanandam V, Khoo A, Geraldes R, Chinthapalli K, Boyd E, Tuzlali H, Price G, Christofi G, Morrow J, McNamara P, McLoughlin B, Lim ST, Mehta PR, Levee V, Keddie S, Yong W, Trip SA, Foulkes AJM, Hotton G, Miller TD, Everitt AD, Carswell C, Davies NWS, Yoong M, Attwell D, Sreedharan J, Silber E, Schott JM, Chandratheva A, Perry RJ, Simister R, Checkley A, Longley N, Farmer SF, Carletti F, Houlihan C, Thom M, Lunn MP, Spillane J, Howard R, Vincent A, Werring DJ, Hoskote C, Jager HR, Manji H, Zandi MS. The emerging spectrum of COVID-19 neurology: clinical, radiological and laboratory findings. Brain. 2020 Oct 1;143(10):3104-3120. doi: 10.1093/brain/awaa240. PMID 32637987
- [Result] Scherlinger M, Felten R, Gallais F, Nazon C, Chatelus E, Pijnenburg L, Mengin A, Gras A, Vidailhet P, Arnould-Michel R, Bibi-Triki S, Carapito R, Trouillet-Assant S, Perret M, Belot A, Bahram S, Arnaud L, Gottenberg JE, Fafi-Kremer S, Sibilia J. Refining "Long-COVID" by a Prospective Multimodal Evaluation of Patients with Long-Term Symptoms Attributed to SARS-CoV-2 Infection. Infect Dis Ther. 2021 Sep;10(3):1747-1763. doi: 10.1007/s40121-021-00484-w. Epub 2021 Jul 10. PMID 34245450
- [Result] Tran VT, Riveros C, Clepier B, Desvarieux M, Collet C, Yordanov Y, Ravaud P. Development and Validation of the Long Coronavirus Disease (COVID) Symptom and Impact Tools: A Set of Patient-Reported Instruments Constructed From Patients' Lived Experience. Clin Infect Dis. 2022 Jan 29;74(2):278-287. doi: 10.1093/cid/ciab352. PMID 33912905
- [Result] Townsend L, Dowds J, O'Brien K, Sheill G, Dyer AH, O'Kelly B, Hynes JP, Mooney A, Dunne J, Ni Cheallaigh C, O'Farrelly C, Bourke NM, Conlon N, Martin-Loeches I, Bergin C, Nadarajan P, Bannan C. Persistent Poor Health after COVID-19 Is Not Associated with Respiratory Complications or Initial Disease Severity. Ann Am Thorac Soc. 2021 Jun;18(6):997-1003. doi: 10.1513/AnnalsATS.202009-1175OC. PMID 33413026